CLINICAL TRIAL: NCT04293393
Title: Phase II, Randomized, Open-label, International, Multicenter Study to Compare Efficacy of Standard Chemotherapy vs. Letrozole Plus Abemaciclib as Neoadjuvant Therapy in HR-positive/HER2-negative High/Intermediate Risk Breast Cancer Patients
Brief Title: Neoadjuvant Study Chemotherapy vs Letrozole + Abemaciclib in HR+/HER2- High/Intermediate Risk Breast Cancer Patients
Acronym: CARABELA
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Spanish Breast Cancer Research Group (Other)
Collaborators: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GEICAM/2019-01; 2019-002123-15 (EudraCT Number)
Record Dates: First submitted 2020-02-28; First posted 2020-03-03 (Actual); Last update posted 2025-09-19 (Actual); Status verified 2025-09

CONDITIONS: Early Breast Cancer
Keywords: Abemaciclib; Neoadjuvant; HR positive; HER2 negative; High/intermediate risk
MeSH Terms: conditions — Breast Neoplasms | interventions — Doxorubicin; liposomal doxorubicin; Cyclophosphamide; taxane; Paclitaxel; Docetaxel; Letrozole; abemaciclib; Gonadotropin-Releasing Hormone; Goserelin; Leuprolide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm A: Doxorubicin plus cyclophosphamide and taxane (Active Comparator): Doxorubicin 60mg/m2 and cyclophosphamide 600mg/m2 (AC) every 21 days for 4 cycles followed by weekly paclitaxel 80mg/m2 for 12 weeks or 3-weekly docetaxel 100mg/m2 for 4 cycles.
  Approximately duration of 24 weeks (6 months).
  Interventions: Drug: Doxorubicin; Drug: Cyclophosphamide; Drug: Taxane
- Arm B: Letrozole plus abemaciclib +/- LHRH (Experimental): Letrozole 2.5mg orally daily + abemaciclib 150mg orally every 12 hours on a continuous dosing schedule, +/- luteinizing hormone-releasing hormone (LHRH) analogs in premenopausal women, up to 12 months, in 28-day cycles.
  Interventions: Drug: Letrozole; Drug: Abemaciclib; Drug: LHRH Analogue

INTERVENTIONS:
Drug: Doxorubicin — Doxorubicin 60mg/m2 and cyclophosphamide 600mg/m2 (AC) every 21 days for 4 cycles followed by weekly paclitaxel 80mg/m2 for 12 weeks or 3-weekly docetaxel 100mg/m2 for 4 cycles.
  Other Names: Caelyx
  Arms: Arm A: Doxorubicin plus cyclophosphamide and taxane
Drug: Cyclophosphamide — Doxorubicin 60mg/m2 and cyclophosphamide 600mg/m2 (AC) every 21 days for 4 cycles followed by weekly paclitaxel 80mg/m2 for 12 weeks or 3-weekly docetaxel 100mg/m2 for 4 cycles.
  Other Names: Genoxal
  Arms: Arm A: Doxorubicin plus cyclophosphamide and taxane
Drug: Taxane — Doxorubicin 60mg/m2 and cyclophosphamide 600mg/m2 (AC) every 21 days for 4 cycles followed by weekly paclitaxel 80mg/m2 for 12 weeks or 3-weekly docetaxel 100mg/m2 for 4 cycles.
  Other Names: Paclitaxel; Docetaxel
  Arms: Arm A: Doxorubicin plus cyclophosphamide and taxane
Drug: Letrozole — Letrozole 2.5mg orally daily + abemaciclib 150mg orally every 12 hours on a continuous dosing schedule, +/- LHRH analogs in premenopausal women, up to 12 months, in 28-day cycles
  Other Names: Femara
  Arms: Arm B: Letrozole plus abemaciclib +/- LHRH
Drug: Abemaciclib — Letrozole 2.5mg orally daily + abemaciclib 150mg orally every 12 hours on a continuous dosing schedule, +/- LHRH analogs in premenopausal women, up to 12 months, in 28-day cycles
  Other Names: Verzenios
  Arms: Arm B: Letrozole plus abemaciclib +/- LHRH
Drug: LHRH Analogue — Letrozole 2.5mg orally daily + abemaciclib 150mg orally every 12 hours on a continuous dosing schedule, +/- LHRH analogs in premenopausal women, up to 12 months, in 28-day cycles
  Other Names: Goserelin; Leuprolide
  Arms: Arm B: Letrozole plus abemaciclib +/- LHRH

SUMMARY:
Phase II, randomized, open-label, international, multicenter study to compare efficacy of standard chemotherapy vs. letrozole plus abemaciclib as neoadjuvant therapy in HR-positive/HER2-negative high/intermediate risk breast cancer patients

DETAILED DESCRIPTION:
This is an international, multicenter, open-label, randomized phase II study in the neoadjuvant setting.

Approximately 200 premenopausal and postmenopausal women with Hormone Receptor (HR)-positive/Human Epidermal Growth Factor Receptor 2 (HER2) negative Breast Cancer (BC) of intermediate/high risk determined by Ki67 index ≥ 20% on untreated breast tissue and centrally assessed, with indication of neoadjuvant treatment, will be included. Patients with Early Breast Cancer (EBC) on stages II-III (tumor size (T) > 2cm - T3, T4b, and lymph node involvement (N) N0-2) according to the 8th edition of the Union for International Cancer Control (UICC) TNM Classification. The subgroup with tumors T2 N0 will include high risk patients based on Ki67 index > 30% or Ki67 index between 20% and 30% and Progesterone Receptor (PgR) negative and/or histological grade 3.

Patients will be stratified according to the disease stage (II vs. III), menopausal status (premenopausal vs. postmenopausal) and Ki67 index (Ki67 < 30% vs. Ki67 ≥ 30%).

Once the screening process (locally at site and at the central laboratory) is completed, fully eligible patients will be randomized in a 1:1 fashion to the control arm with standard Chemotherapy (CT) based on anthracyclines and taxanes or to the experimental arm with letrozole + abemaciclib.

All patients will be treated according to the stipulations below, unless any of the following occur: unacceptable toxicity, progressive disease, or withdrawal of informed consent, whatever occurs first.

After the last dose of any of the drugs in the neoadjuvant combinations, in both treatment arms definitive surgery will be performed. For Arm A not earlier than 21 days and not later than 42 days after the last dose of chemotherapy, and for Arm B within 7 days from the last dose of abemaciclib and/or letrozole, unless toxicities are not recovered completely in any treatment arm.

ELIGIBILITY:
Inclusion Criteria:

Patients are eligible to be enrolled in the study only if they meet all of the following criteria:

1. Written informed consent prior to any specific study procedures.
2. Women ≥ 18 years of age.
3. Documentation of histologically confirmed primary invasive adenocarcinoma of the breast.
4. Availability of a primary tumor tissue sample obtained during the diagnostic process before treatment for the central assessment of Ki67 index.
5. Documentation of Hormone Receptor (HR) positive and Human Epidermal Growth Factor Receptor 2 (HER2) negative Breast Cancer (BC) based on local laboratory determination.

   * HR positive is defined as more than or equal to 10% positive cells by Immunohistochemistry (IHC) for ER and/or progesterone receptor (PgR).
   * HER2 negative tumor is determined according to recommendations of American Society of Clinical Oncology/College of American Pathologists (ASCO/CAP) 2018 guidelines.
6. Intermediate and high risk patients based on Ki67 index value (≥ 20%) determined at a central laboratory.
7. Patients should be in the following clinical stages of disease according to the 8th edition of the TNM Classification of Breast Cancer by the Union for International Cancer Control (UICC): T2 (> 2cm) - T3, T4b, N0 - N2, M0 (stages IIA, IIB, IIIA or IIIB). Subpopulation with tumors T2 N0 M0 will include high risk patients based on Ki67 index > 30% or Ki67 index between 20-30% and PgR negative with or without histological grade 3.
8. Patients diagnosed with multifocal or multicentric breast cancer will be eligible for the study if only 2 tumor lesions have been confirmed in the clinical evaluation and both lesions comply with the characteristics required by the protocol (please, refer to previous inclusion criteria).
9. Indication of neoadjuvant treatment.
10. At the time of presentation, patients must be candidates for potentially curative surgery by surgeon's assessment.
11. Sentinel lymph node biopsy (SLNB) will be preferable after the neoadjuvant treatment. Those patients with SLNB before the neoadjuvant treatment will be eligible for the study only if the SLNB has a negative result (N0). One Step Nucleic Acid Amplification (OSNA) method is not allowed.
12. Premenopausal and postmenopausal women. Postmenopausal status is defined as:

    * Patient underwent bilateral oophorectomy, or
    * Age ≥ 60 years, or
    * Age < 60 years and amenorrhea for 12 or more months (in the absence of chemotherapy, tamoxifen, toremifene or ovarian suppression) and Folliculostimulating hormone (FSH) and plasma estradiol are in the postmenopausal ranges per local normal ranges.

    All women who do not meet the criteria for postmenopausal status are considered premenopausal for the purpose of this trial.
13. Eastern Cooperative Oncology Group (ECOG) performance status (PS) of 0 or 1.
14. Patients are able to swallow oral medications.
15. Adequate organ and bone marrow function:

    * Absolute neutrophil count (ANC) ≥ 1,500/mm3 (1.5x109/L);
    * Platelets ≥ 100,000/mm3 (100x109/L);
    * Hemoglobin (Hgb) ≥ 8g/dL (80g/L) (erythrocyte transfusions are permitted; initial treatment must not begin earlier than the day after the erythrocyte transfusion);
    * Total serum bilirubin ≤ 1.5x Upper Limit of Normal (ULN) (≤ 2x ULN and direct bilirubin within normal limits if Gilbert´s disease);
    * Aspartate aminotransferase (AST) and Alanine aminotransferase (ALT) ≤ 3x ULN.
16. Left ventricular ejection fraction (LVEF) ≥ 50% measured by multiple-gated acquisition scan (MUGA) or echocardiogram (ECHO).
17. For premenopausal women: agreement to remain abstinent or use single or combined non-hormonal contraceptive methods that result in a failure rate of < 1% per year during the treatment period and for at least 3 weeks after the last dose of study treatment. Abstinence is only acceptable if it is in line with the preferred and usual lifestyle of the patient. Periodic abstinence (e.g., calendar, ovulation, symptothermal, or post-ovulation methods) and withdrawal are not acceptable methods of contraception. Examples of non-hormonal contraceptive methods with a failure rate of < 1% per year include tubal ligation, male sterilization, and certain intrauterine devices. Alternatively, two methods (e.g., two barrier methods such as a condom and a cervical cap) may be combined to achieve a failure rate of < 1% per year. Barrier methods must always be supplemented with the use of a spermicide.
18. Negative serum pregnancy test within 7 days of the first dose of abemaciclib for premenopausal women, and for women who have experienced menopause onset < 12 months prior to first dose of therapy.
19. Patients consent to biological sample provision for biomarker exploratory analyses.
20. Willingness and ability to comply with scheduled visits, treatment plan, laboratory tests and other study procedures.

Exclusion Criteria:

Patients will be excluded from the study if they meet any of the following criteria:

1. Previous anti-cancer treatment with therapeutic intent for current breast cancer is not allowed.
2. Inflammatory breast cancer, multifocal/multicentric breast cancer with ≥ 3 tumor lesions or synchronous bilateral invasive breast cancers are not eligible.
3. Serious and/or uncontrolled preexisting medical condition(s) that, in the judgment of the investigator, would preclude participation in this study (for example, interstitial lung disease, severe dyspnea at rest or requiring oxygen therapy, severe renal impairment [e.g. estimated creatinine clearance < 30ml/min], history of major surgical resection involving the stomach or small bowel, or preexisting Crohn's disease or ulcerative colitis or a preexisting chronic condition resulting in baseline Grade 2 or higher diarrhea).
4. Patients with rare hereditary problems of galactose intolerance, total lactase deficiency or glucose- galactose malabsorption.
5. Females who are pregnant or lactating.
6. Active systemic bacterial infection (requiring intravenous [IV] antibiotics at time of initiating study treatment), fungal infection, or detectable viral infection (such as known human immunodeficiency virus positivity or with known active hepatitis B or C [for example, hepatitis B surface antigen positive]. Screening is not required for enrollment.
7. Personal history of any of the following conditions: syncope of cardiovascular etiology, ventricular arrhythmia of pathological origin (including, but not limited to, ventricular tachycardia and ventricular fibrillation), or sudden cardiac arrest.
8. Diagnosis of any other malignancy within 5 years prior to randomization, except for adequately treated basal cell or squamous cell skin cancer, or carcinoma in situ of the cervix or colorectal.
9. Prior hematopoietic stem cell or bone marrow transplantation.
10. Other severe acute or chronic medical or psychiatric condition or laboratory abnormality that may increase the risk associated with study participation or investigational product administration or may interfere with the interpretation of study results and, in the judgment of the investigator, would make the patient inappropriate for entry into this study.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2020-10-02 (Actual); Primary Completion 2023-06-21 (Actual); Study Completion 2033-02-28 (Estimated)

PRIMARY OUTCOMES:
Residual Cancer Burden (RCB) 0-I rate | 24 weeks
  Evaluation of the number of patients with a Residual Cancer Burden (RCB) 0-I index as a measure of efficacy. RCB is a continuous variable derived from the primary tumor dimensions, cellularity of the tumor bed, and axillary nodal burden. It is estimated from routine pathological sections of the primary breast tumor site and the regional lymph nodes after the completion of Neoadjuvant therapy. The pathological variables include bidimensional diameters of the primary tumor bed, the proportion of primary tumor area containing invasive carcinoma, the number of positive lymph nodes, and the diameter of the largest nodal metastasis

SECONDARY OUTCOMES:
Changes in Ki67 index value | 2 weeks
  The percentage of decrease in the geometric mean of Ki67 index value after 2 weeks of treatment in both treatments arms.
  Number of patients with cell cycle arrest (Ki67 < 2.7%) after 2 weeks of treatment in both treatment arms.
RCB 0+I versus RCB-II versus RCB-III | 24 weeks
  RCB is classified in four classes based on the residual disease (RD):
  * RCB-0 defined as pathological complete response.
  * RCB-I defined as minimal RD.
  * RCB-II defined as moderate RD.
  * RCB-III defined as extensive RD.
Rate of Preoperative Endocrine Prognostic Index (PEPI) score 0 at surgery in both treatment arms | 24 weeks
  PEPI requires pathological stage (tumor size and nodal status), level of Ki67 protein, and Allred ER score measured on the surgical specimen. PEPI score 0 includes pT1 or pT2, pN0, Ki67 ≤ 2.7%, Allred score > 2
Clinical response measured by magnetic resonance imaging (MRI) | 24 weeks
  According to RECIST v1.1 in both treatment arms. Clinical Response Rate (CRR) is defined as the proportion of subjects with complete or partial radiographic response. Complete Response (CR) and Partial Response (PR) definitions are assessed by MRI at baseline and prior to breast surgery, with or without regional lymph nodes surgery, and categorized according to percent reduction in tumor size.
Rate of breast conservative surgery (BCS) in both treatment arms. | 24 weeks
  Rate of breast conservative surgery (BCS): defined as the proportion of patients who achieved breast-conserving surgery between both treatment arms.
iEFS (invasive Event Free Survival) in both treatment arms. | Up to 10 years
  Invasive event free survival (iEFS): defined as time from randomization to progressive disease or invasive disease recurrence (local, regional, distant, or contralateral), or death from any cause. Invasive disease recurrence is defined as:
  * Ipsilateral invasive breast tumor recurrence (including second primary invasive breast cancer): an invasive breast cancer involving the same breast parenchyma as the original primary lesion.
  * Ipsilateral regional invasive breast cancer recurrence (i.e., an invasive breast cancer in the axilla, other regional lymph nodes, chest wall, and/or skin of the ipsilateral breast).
  * Distant recurrence (i.e., evidence of breast cancer in any anatomic site outside local and/or regional location and that has been either histologically confirmed or clinically diagnosed as recurrent invasive breast cancer)
  * Contralateral invasive breast cancer
  * Second primary invasive cancer of non-breast origin.
Number of patients with adverse events | 24 weeks
  Safety will be assessed by standard clinical and laboratory tests (haematology, serum chemistry). Adverse Events (AEs) grade will be defined by the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) version 5.0. AEs terms will be coded according to MedDRA dictionary.
To assess molecular downstaging for high risk genomic groups defined by a multigene expression panel. | 24 weeks
  Gene expression data provided by a multigene expression panel in sequential tumor biopsies.

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Hospital General Universitario Gregorio Marañon; Study Director, Study Director — Hospital Universitario Virgen de la Victoria; Study Director, Study Director — Instituto Valenciano de Oncología
Locations (28):
- Spain (28):
  - Complejo Hospitalario Universitario de Santiago (CHUS), Santiago de Compostela, A Coruña
  - Institut Català d'Oncología (ICO) L'Hospitalet, L'Hospitalet de Llobregat, Barcelona
  - Hospital Universitario Marqués de Valdecilla, Santander, Cantabria
  - Consorcio Hospitalario Provincial de Castellón, Castellon, Castelló
  - Hospital Universitario Donostia, San Sebastián, Donostia
  - Hospital Álvaro Cunqueiro, Vigo, Pontevedra
  - Complejo Hospitalario Universitario A Coruña (CHUAC), A Coruña
  - Hospital General Universitario de Alicante, Alicante
  - Hospital Universitario de Badajoz, Badajoz
  - Hospital Universitario de Burgos, Burgos
  - Hospital Universitario San Pedro de Alcántara, Cáceres
  - Hospital Universitario Reina Sofía, Córdoba
  - Institut Català d'Oncología (ICO) Girona, Girona
  - Complejo Hospitalario de Jaén, Jaén
  - Hospital General Universitario Gregorio Marañón, Madrid
  - Hospital Universitario Ramón y Cajal, Madrid
  - Hospital Clínico San Carlos, Madrid
  - Hospital Clínico Universitario Virgen de la Victoria, Málaga
  - Hospital General Universitario Morales Meseguer, Murcia
  - Hospital Universitario Nuestra Señora de Candelaria, Santa Cruz de Tenerife
  - Hospital Universitario Virgen del Rocío, Seville
  - Hospital Virgen de la Salud, Toledo
  - Fundación Instituto Valenciano de Oncología (FIVO), Valencia
  - Hospital Clínico Universitario de Valencia, Valencia
  - Hospital Universitari i Politécnic La Fe, Valencia
  - Hospital Universitario Reina Sofía, Valencia
  - Hospital Clínico Universitario Lozano Blesa, Zaragoza
  - Hospital Universitario Miguel Servet, Zaragoza

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Spanish Breast Cancer Research Group (GEICAM) is a Spanish Breast Cancer Research Group — http://www.geicam.org